CLINICAL TRIAL: NCT01171079
Title: Use of an Oxidized Regenerated Cellulose After Thyroid Surgery: A Prospective, Randomized Study
Acronym: ORC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Other Study IDs: ORC-100
Record Dates: First submitted 2010-07-26; First posted 2010-07-28 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Thyroidectomy
Keywords: postoperative adhesion after thyroidectomy

ARMS (1):
- Interceed (Experimental)
  Interventions: Device: application of oxidized regenerated cellulose

INTERVENTIONS:
Device: application of oxidized regenerated cellulose

SUMMARY:
The purpose of this study is to evaluate the effects and safety of oxidized, regenerated cellulose as an absorbable adhesion barrier after thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* operable thyroid neoplasm

Exclusion Criteria:

* a history of previous neck surgeries or uncontrolled medical diseases such as hyperthyroidism, diabetes, and hypertension
* administration of non-steroidal anti-inflammatory drugs (NSAIDs) or anti-platelet agents within 1 week before surgery

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Yigit O, Uslu Coskun B, Coskun H, Yilmaz B, Alkan S, Cinar U, Dadas B. Efficacy of anti-adhesive barriers in secondary thyroidectomy: an experimental study. Laryngoscope. 2004 Sep;114(9):1668-73. doi: 10.1097/00005537-200409000-00031. PMID 15475802
- [Background] Yilmaz O, Genc A, Taneli F, Demireli P, Deliaga H, Taneli C. Assessment of the efficacy of absorbable adhesion barriers on dissection in esophagus operations. Int J Pediatr Otorhinolaryngol. 2007 Mar;71(3):409-14. doi: 10.1016/j.ijporl.2006.11.010. Epub 2006 Dec 11. PMID 17161874